CLINICAL TRIAL: NCT04083508
Title: A Clinical Study to Assess the Feasibility of a Controlled Human Plasmodium Vivax Malaria Infection Model Through Sporozoite Infection in Thai Adults
Brief Title: Vivax Malaria Human Infection Studies in Thailand
Acronym: MIST1
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: Mahidol University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MAL19002
Record Dates: First submitted 2019-09-05; First posted 2019-09-10 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Plasmodium Vivax Infection

STUDY DESIGN:
Intervention Model Description: Mosquito-bite controlled human challenge infection
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Malaria challenge (Experimental): Malaria Sporozoite Challenge by mosquito bites.
  Interventions: Other: Mosquito bites

INTERVENTIONS:
Other: Mosquito bites — Successful feeding of 5 infected P. vivax mosquitoes

SUMMARY:
This study is a human challenge study to assess the feasibility and safety of controlled human malaria infection (via P. vivax sporozites) in healthy volunteers, and to develop a bank of P. vivax-infected blood for use in future controlled human P. vivax malaria infection studies. Additional objectives are to obtain data on host immune response to P. vivax infection and pre-treatment gametocytaemia.

This study is funded by the UK Wellcome Trust. The grant reference number are Oxford/MORU: 212336/Z/18/Z and 212336/Z/18/A, and Mahidol University: 212336/A/18/Z and 212336/A/18/A.

DETAILED DESCRIPTION:
Six healthy, malaria-naïve Thai adults, aged between 20 and 55 years will be recruited at the Medical Therapeutics Unit (MTU) in the Hospital for Tropical Medicine, Faculty of Tropical Medicine, Mahidol University, Bangkok. The overall period of participation will be 15 months: a 3-month screening process prior to the Day 0 challenge, followed by 1 year after challenge. All inclusion and exclusion criteria will be checked to ensure eligibility criteria have been met prior to Day 0.

Volunteers will be admitted as inpatients to the CTU on Day -1 ( a day prior to the challenge day). Challenge (bites from 5 infected mosquitoes) will be administered at the Insectarium unit, Department of Entomology, Faculty of Tropical Medicine, Mahidol University. The infected mosquitoes will be prepared by the Malaria Vivax Research unit (MVRU, Faculty of Tropical Medicine, Mahidol University). Following successful feeding by the infectious mosquitoes, volunteers will be monitored daily as inpatients for parasitemia and clinical presentation of malaria infection (Days 1-5).

Beginning on Day 6, volunteers will be assessed twice a day and, at a timepoint that will depend upon the level of parasitaemia and/or degree of the volunteer's symptoms, up to 250 mL of blood will be drawn and then antimalarial treatment will be prescribed. The standard malaria radical cure according to standardguideline will be chloroquine, followed by direct observed of oral primaquine (PQ) 30 mg once daily until a total dose of 10 mg/kg is achieved. Upon confirmation of clinical recovery, completion of chloroquine treatment and laboratory absence of infection, volunteers will be discharged and followed daily as outpatients through completion of oral primoquine therapy.

After completion of antimalarial therapy, all volunteers will continue to be followed for 1 year after Day 0:

* Outpatient CTU visits on Days 28,60, 90, 180, and 365 post-challenge. Procedures to be performed during these visits will include review of symptom diary cards, medical history, physical examination and assessment of adverse events. Blood samples will also be obtained to detect malaria antigens and assess immune response.
* Volunteers will be contacted by study staff every 2 weeks between visits until Day 365, to inquire for malaria symptoms or other adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult aged 20 to 55 years with weight more than 50 kg.
* Blood group O.
* Red blood cells positive for the Duffy antigen/chemokine receptor (DARC).
* CYP2D6 alleles consistent with normal metaboliser status
* Normal blood levels of Glucose-6-phosphate dehydrogenase (G6PDH) by the WHO definition.
* COVID-19 vaccination at least two doses of COVID-19 vaccine(s) approved by WHO.
* Agree to practice continuous effective contraception for the duration of study period until 3 months post-challenge.
* Agreement to refrain from blood donation during the course of the study and for 1 year after the end of their involvement in the study.
* Willing to take a curative antimalarial regimen following challenge.
* Willing to be admitted in the Hospital for Tropical Diseases for blood donation and clinical monitoring, until antimalarial treatment is completed and their symptoms are settling.
* Willing to reside in Bangkok for the duration of the study, until all antimalarial treatment has been completed.
* Reachable (24/7) by mobile phone during the period between challenge CHMI and completion of all antimalarial treatment.
* Able to read and write in Thai and able to answer ALL questions on the informed consent questionnaire correctly.
* Provided written informed consent to participate in the trial.
* Educational level: has at least an undergraduate degree.
* Cardiovascular risk assessment is low (less than 10% in the next 10 years according to the cardiovascular risk assessment from Thai NCD Division, DDC, MoPH (2016)

Exclusion Criteria:

* History of clinical malaria.
* Positive malaria PCR OR malaria film OR malaria serology (recent exposure)
* History of severe allergy to mosquito bite
* Presence of any medical condition (either physical or psychological) which in the judgment of the investigator would place the participant at undue risk or interfere with the results of the study (e.g. serious underlying cardiac, renal, hepatic or neurological disease; severe malnutrition; congenital defects or febrile condition)
* Presence of chronic disease or chronically use of medication.
* Plan to travel outside of Bangkok within the period of challenge until 3 months after.
* Use of systemic antibiotics with known antimalarial activity in the 30 days before challenge (e.g. trimethoprim-sulfamethoxazole, doxycycline, tetracycline, clindamycin, erythromycin, fluoroquinolones and azithromycin).
* Use of immunoglobulins or blood products (e.g. blood transfusion) at any time in the 1 year preceding enrolment.
* Venipuncture unlikely to allow blood donation according to the protocol as determined by the investigator.
* Receipt of an investigational product or any vaccine in the 30 days preceding enrolment (D0), or planned receipt during the study period.
* Prior receipt of an investigational vaccine likely to impact on interpretation of the trial data or the P. vivax parasite as assessed by the Investigator.
* Any confirmed or suspected immunosuppressive or immunodeficient state, including HIV infection, asplenia, history of splenectomy, recurrent, severe infections, and chronic infection.
* Immunosuppressant medication within the past 6 months preceding enrolment (D0) (inhaled and topical steroids are allowed).
* History of allergic disease or reactions likely to be exacerbated by malaria infection.
* Female participant who is pregnant, lactating or planning pregnancy during the course of the study.
* Contraindications to the use of antimalarial treatment (e.g. chloroquine or primaquine or atovaquone / proguanil, DHA piperaquine).
* Use of medications known to have a potentially clinically significant interaction with antimalarial drug that will be used in this study (chloroquine or primaquine or atovaquone / proguanil, DHA/ piperaquine).
* Use of medications known to cause prolongation of the QT interval as state in the section of prohibited drugs that may have effect on prolongation of the QT interval.
* Known existing positive family history in both 1st AND 2nd degree relatives < 50 years old for cardiac disease.
* Family history of congenital QT prolongation or sudden death.
* Any clinical condition known to prolong the QT interval.
* History of cardiac arrhythmia, including clinically relevant bradycardia.
* Screening ECG demonstrates a QTc interval ≥ 450 ms
* Suspected or known or history of alcohol abuse
* Suspected or known or history of drug abuse.
* Concurrently participating in another clinical study, at any time during the study period.
* Haemoglobin < 13 g/dL in male, < 12g/dL in female (Thai Red Cross).
* Finding on safety laboratory values as defined below:
* AST > 40 U/L for male, and > 32 U/L for female (upper normal range), or
* ALT > 41 U/L for male, and > 33 U/L for female (upper normal range), or
* Total Bilirubin > 1.2 mg/dL, (upper normal range), or
* Creatinine (Cr) > 1.17 mg/dL for male, and > 0.95 mg/dL for female (upper normal range), or
* Abnormalities corrected calcium and magnesium blood levels, or
* Fasting blood sugar (FBS) > 100 mg/dL
* Thalassaemia disease or haemoglobinopathies.
* Positive for a blood borne or vector borne infectious disease (HIVI-II, HBV, HCV, Dengue, Zika, Chikungunya, Filariasis, JE, and malaria antigen, Anti HTLVI and Anti-HTLVII antibody, Syphilis test (TPHA)
* Positive for COVID-19 testing as diagnosed by RT-PCR

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Estimated)
Dates: Start 2020-10-05 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Successful infection of controlled P. vivax sporozoite human challenge | up to 21 days after challenge
  Measured by successful infection (development of detectable persistent parasitaemia) and malaria clinical symptoms, if any, after mosquito bite malaria sporozoite challenge
(Serious) Adverse Event(s) occurrences of controlled P. vivax sporozoite human challenge | up to 90 days after challenge
  Measured by (S)AE(s) occurrences after mosquito bite malaria sporozoite challenge.
Collection and freezing down of up to 250 mL P. vivax-infected blood from each of the 6 volunteers. | up to 21 days after challenge
  measured by successful collection and freezing down of up to 250 mL P. vivax-infected blood from each of the 6 volunteers.

SECONDARY OUTCOMES:
Cellular Immune response to primary P. vivax infection. | up to 1 year after challenge
  immune cells including Innate and adaptive immune cells react and express during the PV infection (profile and frequency)
Humoral Immune response to primary P. vivax infection. | up to 1 year after challenge
  Immune cells defense PV antigen by determining the level of antibody response and inflammatory cytokine
Gametocytaemia following primary P. vivax infection delivered by the mosquito bite | up to 1 year after challenge
  Gametocyte qPCR following primary P. vivax infection delivered by the mosquito bite

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Day, MD, Principal Investigator — University of Oxford
Locations (1):
- Faculty of Tropical Medicine, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: Yes
With participant's consent, suitably anonymised clinical data and results from blood analyses stored in the database may be shared according to the terms defined in the MORU data sharing policy with other researchers to use in the future.
Time Frame: After completion of trial activities and reporting
URL: https://www.tropmedres.ac/units/moru-bangkok/bioethics-engagement/data-sharing

REFERENCES:
- [Derived] Naemiratch B, Kulpijit N, Ruangkajorn S, Day NPJ, Prachumsri J, Cheah PY. Experiences, perceptions and ethical considerations of the malaria infection study in Thailand. BMC Med Ethics. 2025 Jan 28;26(1):14. doi: 10.1186/s12910-024-01160-7. PMID 39875955

DOCUMENTS (2):
  • Study Protocol (2022-02-14): https://cdn.clinicaltrials.gov/large-docs/08/NCT04083508/Prot_002.pdf
  • Statistical Analysis Plan (2021-05-10): https://cdn.clinicaltrials.gov/large-docs/08/NCT04083508/SAP_001.pdf